CLINICAL TRIAL: NCT04619836
Title: Cost-effectiveness of the Care Pathways - Effects of Patient Segmentation to Quality and Costs of Type 2 Diabetes and Substance Abuse Care and Services
Brief Title: Cost-effectiveness of the Care Pathways
Status: Enrolling by invitation | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R19134
Record Dates: First submitted 2020-06-26; First posted 2020-11-06 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabete Type 2; Substance Abuse
Keywords: patient segmentation; effectiveness; cost-effectiveness; quality of life; quality of care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- segmentation type 2 diabetes patitents: Those type 2 diabetes patients, who have segmenteted for four groups to organinize cervices and self care
- Non-segmentation type 2 diabetes patients: Those type 2 diabetes patiets who have not segementated
- Segmentation substance abuse clients: Those type substance abuse clients, who have segmenteted for four groups to organinize cervices and self care
- Non-segmentation substance abuse clients: Those type substance abuse clients, who have not segmenteted

SUMMARY:
In this study we research patient segmentation made by Suuntima-service and it´s impacts to Quality of care, Service use and Costs of care among Type 2 Diabetes patients and Substance Abuse patients.

With this Suuntima-servise based segmentation we assume to find appropriate services and Self-Management to allocate Type 2 Diabetes and Substance Abuse patients. We plan their care pathways by Suuntiman-service customership strategies (Self-acting, community, co-operation, network).

DETAILED DESCRIPTION:
The study recruits 270 adult-type diabetics and 200 clients of substance abuse services for each of the four client segments (self-employment, community, cooperation, network client) and the comparison group.

Based on previous evaluations and studies of the Suuntima service, it is assumed that there will be 60% self-acting customers, 20% community customers, 10% co-operation customers, 10% network customers, therefore patients must be recruited sample. Thus, a total of about 1,350 to 1,500 patients are recruited for adult-type diabetes patients, and 1,000 to 1,200 clients for substance abuse services until sufficient representation is obtained for each clientele.

Every adult patients with type 2 diabetes who are admitted to the caregiver's preparatory diabetic nurse appointment for the annual diabetes control will be asked to participate in the study until the number of patients required for the study has been accumulated. With regard to the substance abuse process, all clients who come to the substance abuse nurse's office are asked to participate in the study.

Nursing staff review the information document with the subjects in an understandable way and the subjects are given the opportunity to ask questions about the study. If they choose to participate in the study, they will be asked to comply with consent to participate in the study.A Suuntima is made for the research subject and the customership and the type of use of the services, ie the servicepath, are defined. At the beginning, the research patients fill in a 15D questionnaire measuring the quality of life and a service experience meter (NPS, Net Promoter Score) and answer questions about height, weight, smoking habbits and how they manages in their everyday life. Clients of substance abuse services answer also questions about substance use. To monitor the quality and effectiveness of treatment, clinical variables are collected from the patient information system according to the recommendation of the National Diabetes Treatment Quality Register (Glucose hemoglobin, LDL cholesterol, albumin-creatinine ratio). Similarly, the necessary clinical parameters (serum glutamyltransferase (GT), serum low-carbohydrate transferrin (CDT), and drug screen) are collected from clients of substance abuse to monitor the quality and effectiveness of treatment.

In addition, the study collects information on the use of the health and social services and costs in general, as well as on the use and costs of services related to diabetes or substance abuse are collected from the patient information systems of both the health centers and Tampere Univercity hospital information systems of municipal social services. Laboratory data are collected from Fimlab's information systems with the permission of the registrar, and cost data for specialist care are collected from Tays' Mynla system.

Follow-up data will be collected after one and two years in connection with diabetes monitoring, in which case the above-mentioned data collection will be repeated. For substance abuse clients, monitoring is performed at 6 months and 12 months. In addition, the follow-up visit examines with a questionnaire whether the customer path has been realized as planned during the follow-up period.

In the autumn of 2020, the health care professionals participating in the study will be interviewed about the implementation of customer paths during the year. Interviews are recorded, transcribed. Participation in the interview is voluntary and your information will be collected without any unique identifiers. The information is processed in such a way that no individual interviewee can be directly identified from them.

At the same time, similar information is collected at the reference health centers agreed in Pirkanmaa for adult-type diabetic patients and substance abuse patients, whose services are not planned according to the Suuntima service customership carepathways.

ELIGIBILITY:
Inclusion Criteria:

* every diabetes type 2 patiets, who visit health to center diabetes nurse and substance abuse client who visit health and socialcenter, and whose services and self management are planned by Suuntima segmentation customership srategies

Exclusion Criteria:

* under 18 years, over 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: and
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire (Prom) | 2 years
  change in quality of life measured by 15D- questionnaire
Net promoter score questionnaire (NPS) | 2 years
  effects to NPS questionnaire
Effects to health and social services use | 2 years
  volume of services will be collected from national patient register
Effects to health and social services use | 2 years
  costs of services will be collected from national patient register
Effects to quality of care with laboratory mesurements | 2 years
  glucose hemoglobin (B-HbA1c)
Effects to quality of care with laboratory mesurements | 2 years
  plasma low density lipoprotein cholesterol level (f-P-Kol-LDL-cholesterol)
Effects to quality of care with laboratory mesurements | 2 years
  Urine albumin/creatinine ratio (U-Alb/Krea)
Effects to quality of care with laboratory mesurements | 2 years
  seerum Gamma Glutamyl Transferase (GGT)
Effects to quality of care with laboratory mesurements | 2 years
  carbohydrate deficient transferrin (CDT)
Effects to quality of care with laboratory mesurements | 2 years
  Urine drugtest
Effects to quality of care with physiological mesurements | 2 years
  Weight in kilograms
Effects to quality of care with physiological mesurements | 2 years
  Height in meters
Effects to quality of care with questionnaire | 2 years
  smoking habits questionnaire

SECONDARY OUTCOMES:
How to guide patients | 1 year
  interview to nurses, qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Sari Mäkinen, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere university hospital, Tampere, Finland